CLINICAL TRIAL: NCT00772681
Title: Phase IV Clinical Study Evaluating The Efficacy of Chemoradiotherapy Following Neoadjuvant Treatment With Docetaxel and Cisplatin in Indifferentiated and Non-keratinized Squamous Cell Carcinoma of Nasopharynx
Brief Title: Efficacy of Chemoradiotherapy After Neoadjuvant Cisplatin and Docetaxel in the Nasopharynx Carcinoma
Acronym: Tax-Nazo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976F_6007
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: docetaxel and cisplatin

INTERVENTIONS:
Drug: docetaxel and cisplatin — 3 cycles of docetaxel 75mg/m2 and 100mg/m2 cisplatin combination every 3 weeks

SUMMARY:
* To assess the efficacy of docetaxel, cisplatin combination in terms of disease free survival.
* Time to progression of the disease in terms of local and distant failure; assess the survival time, and assess the objective (clinical and radiological) response rate and the safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed, patients with stage T2b-T4N1 or TanyN2-3 undifferentiated or nonkeratinized squamous cell carcinoma of nasopharynx who are candidate for curative radiotherapy.
* ECOG Performance Status is 0-1
* Weight loss within last 6 months <10% of body weight
* Acceptable haematological profile (as defined by a leukocyte count ≥ 4000/mm3, a platelet count ≥ 100.000mm3 and Hb ≥ 9g/100mL), and adequate renal function (as defined by serum creatinine ≤ 1.5mg/dl), and hepatic function (as defined by bilirubin ≤ 1.5 x maximum normal value even with hepatic metastasis; transaminases (ALT, AST) ≤ 1.5 x maximum normal value; alkaline phosphatase ≤ 2.5 x maximum normal value, except in case of a bone metastasis)

Exclusion Criteria:

* Patients with stage IVC or metastatic disease
* Patients treated with chemotherapy for nasopharyngeal cancer
* Patients treated with radiotherapy to head and neck region
* Concomitant use of another anti-cancer therapy
* Patients treated with amifostine or pilocarpine during protocol treatment.
* Unstable medical condition that makes the patient unable to take part in a clinical study (congestive heart failure, serious arrhythmia, uncontrolled diabetes mellitus), history of myocardial infarction within last 6 months, massive pleural, peritoneal or pericardial effusion; or presence of serious uncontrolled infection.
* Presence of other tumours different from carcinoma of the skin except melanoma and carcinoma in situ of the breast and cervix with disease free survival less than 5 years.
* Pregnancy or breastfeeding. In women of childbearing potential and in men, an adequate contraceptive method must be used
* Social or psychological condition that render the patient inadequate for the follow-up of the study
* Contraindication for any of the study drugs (e.g. history of hypersensitivity to any of the ingredients of the study drugs)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Complete response rate after neoadjuvant chemotherapy | From the start date of the treatment to the date of first documented progression of disease or at least until 2 years follow-up period

SECONDARY OUTCOMES:
Percentage of patients whose is disease controlled locally or regionally | from the start date of the treatment to the date of first documented local or regional tumor progression
Median length of overall survival | time interval from the date of treatment to the date of death or at least until 2 years follow-up period
Median length of disease free survival | time interval from the date of treatment to the date of death or at least until 2 years follow-up period
Percentage of alive patients without metastatis | from the start date of the treatment to the date of first documented distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)